CLINICAL TRIAL: NCT03819582
Title: Visual Performance Following Implantation of a Hydrophobic Aspheric Monofocal Intraocular Lens
Brief Title: Visual Performance With a Hydrophobic Aspheric Monofocal IOL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Dr Phillip J Buckhurst, Associate Head of School for Research, University of Plymouth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17/WM/0181
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraocular lens (Experimental): Subjects implanted with the EyeCee One Intraocular lens
  Interventions: Device: EyeCee One intraocular lens

INTERVENTIONS:
Device: EyeCee One intraocular lens — Hydrophobic aspheric monofocal intraocular lens

SUMMARY:
Artificial lenses, otherwise known as intraocular lenses (IOLs), are used to replace the natural crystalline lens within the eye during cataract or refractive lens surgery. Monofocal IOLs are the traditional IOL type used during cataract surgery. These monofocal IOLs provide excellent distance vision, however spectacles are required for reading and intermediate distance tasks. Monofocal Intraocular lenses are the mainstay of cataract surgery, but with advancing technologies and a wider selection of lenses available, demand for improved outcomes, improved lens design and ease of surgical implantation have increased. The purpose of this study is to assess the visual performance of the EyeCee One monofocal intraocular lens. In addition an assessment of the ease of insertion by the surgeon will be quantified.

DETAILED DESCRIPTION:
Artificial lenses, otherwise known as intraocular lenses (IOLs), are used to replace the natural crystalline lens within the eye during cataract or refractive lens surgery. Monofocal IOLs are the traditional IOL type used during cataract surgery. These monofocal IOLs provide excellent distance vision, however spectacles are required for reading and intermediate distance tasks. There are many different designs of monofocal IOLs, all with their own unique optical properties, however there is little evidence to support which optical design provides the best visual outcome. This research project allows us to assess the visual outcomes of a specific monofocal IOL. It also allows us to assess the ease of use of the lens to the surgeon.

Each subject will be evaluated at two visits following IOL implantation; visit 1 (1 month post implantation), Visit 2 (3 months post implantation).

At both post-operative visits the patient will undergo:

Refraction Uncorrected and best corrected distance and near visual acuity measurement Optical biometry to assess ELP Slit lamp biomicroscopy to assess for post-operative complications

At the time of surgery, the ophthalmic surgeon will complete a questionnaire, detailing lens insertion time and ease of use.

ELIGIBILITY:
Inclusion Criteria:

-Clinically significant Cataract requiring cataract surgery

Exclusion Criteria:

* Amblyopia
* Corneal astigmatism of >1.00D
* Dilated pupil size smaller than 5mm
* Macular pathology
* Glaucoma
* Retinal disease
* Corneal disease
* Abnormal iris
* Pupil deformation
* Any previous corneal or intraocular surgery
* Any patient who had surgical complications will also be excluded from participation in the study.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity early post operative | 1 month post operatively
  Visual acuity measured in LogMAR early post operatively
Visual acuity after 3 months post operatively | 3 months post operatively
  Visual acuity measured in LogMAR measured 3 months post operatively

SECONDARY OUTCOMES:
Ease of use to surgeons | During surgery
  Questionnaire completed by the surgeon to determine the usability of the intraocular lens

CONTACTS AND LOCATIONS:
Locations (1):
- BMI Southend Hospital, Westcliff-on-Sea, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No